CLINICAL TRIAL: NCT00950326
Title: A Comparison of Kneipp Hydrotherapy With Conventional Physiotherapy in the Treatment of Osteoarthritis of the Hip or Knee: Protocol of a Prospective Randomised Controlled Clinical Trial
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kneippsche Stiftungen (Other)
Collaborators: Otto-Schönfisch Foundation/ Bad Wörishofen/ Germany (Unknown)
Responsible Party: Kneippsche Stiftungen/ Bad Wörishofen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSF
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis of the Hip or Knee
Keywords: osteoarthritis; hydrotherapy; affusion; conventional physiotherapy; comparison
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- B1-Physio (Active Comparator): In Group B1, patients will be given physiotherapy of the hip or knee joint three times a week
  Interventions: Procedure: Physiotherapy
- A1 Hydro (Experimental): In this group patients will receive a specific hydrotherapeutic procedure in the form of alternate cold and warm thigh affusions ( pouring on water) which will consist of repeated cold and warm water stimulation of the knee and hip region.
  Interventions: Procedure: Affusion
- C- Hydro & Physiotherapy (Active Comparator): Patients with active osteoarthritis of the hip or knee will receive specific, joint-related hydrotherapy in the form of a (daily) alternate cold and warm thigh affusions as well as joint-specific physiotherapy (three times a week).
  Interventions: Procedure: Affusion/ Physiotherapy

INTERVENTIONS:
Procedure: Physiotherapy — In intervention group B1, patients with osteoarthritis of the hip or knee will receive specific physiotherapy of the affected hip or knee joint three times a week, but without any disease-specific hydrotherapy. Because of the holistic approach of the clinic, however, these patients will still receive hydrotherapy at sites other than the affected joint, for example, alternate cold and warm affusions of the back or an ascending lumbar affusion.
  Arms: B1-Physio
Procedure: Affusion — Patients will receive a specific hydrotherapeutic procedure in the form of alternate cold and warm thigh affusions ( pouring on water) which will consist of repeated cold and warm water stimulation of the knee and hip region (daily). Physiotherapy of other regions, such as the back, is permitted but there will be no specific physiotherapy of the hip or knee joint.
  Arms: A1 Hydro
Procedure: Affusion/ Physiotherapy — Patients with active osteoarthritis of the hip or knee will receive specific, joint-related hydrotherapy in the form of a (daily) alternate cold and warm thigh affusions as well as joint-specific physiotherapy (three times a week).
  Arms: C- Hydro & Physiotherapy

SUMMARY:
The study design consists of a prospective randomised controlled three-armed clinical trial, which will be carried out at a specialist clinic for integrative medicine, to investigate the clinical effects of hydrotherapy on osteoarthritis of the knee or hip joint, in comparison with conventional physiotherapy.

DETAILED DESCRIPTION:
The main aim of this three-armed clinical study will be to determine the effects of hydrotherapy with alternate cold and warm affusions of the thigh in the concomitant treatment of osteoarthritis of the hip or knee. The main outcome measures are pain reduction, improvement in the quality of life, and increased movement in the affected joint.

Research questions

1. Does Kneipp hydrotherapy show a measurable effect in the sense of altered clinical findings in the affected knee or hip joint?
2. How effectively does hydrotherapy influence the clinical parameters of pain, range of movement, and function of the affected joint?
3. How effectively does hydrotherapy affect the secondary outcome measures of quality of life, pain experienced, mood, and blood pressure?
4. Do hydrotherapeutic applications simply provide short-term therapeutic success or are there long-term changes in the clinical findings?
5. Are the clinical effects of hydrotherapy comparable with those of conventional physiotherapy of the affected joint?
6. Are the clinical effects of hydrotherapy used as monotherapy comparable with a combination of hydrotherapy and physiotherapy of the affected joint?
7. Do unwanted effects or side effects occur with hydrotherapy?

This study was designed as a prospective randomised controlled clinical trial with three arms, which is to be carried out at a German clinic specialised in integrative medicine, to investigate the clinical effects of hydrotherapy on osteoarthritis of the knee or hip, as compared with conventional physiotherapy.

To achieve maximum scientific accuracy with respect to randomisation, random distribution, avoidance of selection bias, etc., the independent Department of General Medicine and Primary Care of the University of Leipzig Medical School will function as an external evaluation and testing centre.

The design and concept of this study, as well as its ethical validity, were reviewed and approved by the Ethics Committee of the Bavarian State Chamber of Physicians [Ethikkommission der Bayerischen Landesärztekammer], (Study Number 08032, dated 04.05.2008).

One hundred and eighty patients diagnosed with osteoarthritis of hip or knee will be randomly assigned to one of three intervention groups: hydrotherapy, physiotherapy, and both physiotherapy and hydrotherapy of the affected joint. In the first group, patients will receive Kneipp hydrotherapy daily, with water applied in the form of alternate cold and warm thigh affusions (alternating cold and warm water stimulation is particularly relevant to the knee and hip regions).

Patients in the second group will receive physiotherapy of the hip or knee joint three times a week. Patients in the physiotherapy-hydrotherapy combination group will receive both joint-specific physiotherapy three times a week and alternate cold and warm thigh affusions every day.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Symptomatic osteoarthritis of hip or knee (following the revised criteria of the American College of Rheumatology)
* Willingness to comply with follow-up assessments and treatment
* Ability to understand, read and speak German

Exclusion Criteria:

* Endoprothetic replacement of hip or knee joint
* Inflammatory arthropathy of the hip or the knee
* Acute, hot, red and swollen knee or hip joint (unknown focus)
* Inflammatory system diseases which could interfere with the evaluation of the therapy procedure
* CNS diseases, especially epilepsy
* Anamnesis of deep vein thrombosis in the past 12 months
* Severe lung disease such as e.g. COPD stages GOLD III - GOLD IV
* Heart failure NYHA III - NYHA IV
* Myocardial ischemia with or without intervention within the last 3 months before inpatient admission
* Cancer in advanced stage
* Large skin wounds or inflammatory and ulcerated dermatosis of the legs
* Severe febrile infectious diseases
* Non treated hypertension
* Participation in another clinical study within the past four weeks
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the pain intensity of the affected joint during inpatient care, as assessed by the patient and the investigator | 2 Years

SECONDARY OUTCOMES:
I) Mobility of the affected joint II) Quality of life rating for the patient with osteoarthritis, on the basis of the German version of the Arthritis Impact Measurement Scale (AIMS2) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schencking, MD, Principal Investigator — Head of department, Kneipp-Clinic, Bad Wörishofen
Locations (1):
- Kneipp-Clinic, Bad Wörishofen, Bavaria, Germany

REFERENCES:
- [Background] 1. Buckwalter JA, Saltzman C, Brown T: The impact of osteoarthritis: implications for research. Clin Orthop Relat Res 2004;S6-15. 2. Aigner T, Rose J, Martin J, Buckwalter J: Aging theories of primary osteoarthritis: from epidemiology to molecular biology. Rejuvenation Res 2004;7:134-145. 3. Lohmander LS, Gerhardsson d, V, Rollof J, Nilsson PM, Engstrom G: Incidence of severe knee and hip osteoarthritis in relation to different measures of body mass: a population-based prospective cohort study. Ann Rheum Dis 2009;68:490-496. 4. Bijlsma JW, Knahr K: Strategies for the prevention and management of osteoarthritis of the hip and knee. Best Pract Res Clin Rheumatol 2007;21:59-76. 5. Berman BM, Lao L, Langenberg P, Lee WL, Gilpin AMK, Hochberg M: Effectiveness of Acupuncture as Adjunctive Therapy in Osteoarthritis of the Knee. Ann intern Med. 2004; 141:901-910 6. Leardini G, Mascia MT, Stisi S, Sandri G, Franceschini M: [Sanitary costs of osteoarthritis]. Reumatismo 2001;53:316-322. 7. Solignac M: [COART France 2003 report on new socioeconomic data on osteoarthritis in France]. Presse Med 2004;33:S4-S6. 8. Zochling J, March L, Lapsley H, Cross M, Tribe K, Brooks P: Use of complementary medicines for osteoarthritis--a prospective study. Ann Rheum Dis 2004;63:549-554.
- [Derived] Schencking M, Wilm S, Redaelli M. A comparison of Kneipp hydrotherapy with conventional physiotherapy in the treatment of osteoarthritis: a pilot trial. J Integr Med. 2013 Jan;11(1):17-25. doi: 10.3736/jintegrmed2013004. PMID 23464642
- [Derived] Schencking M, Otto A, Deutsch T, Sandholzer H. A comparison of Kneipp hydrotherapy with conventional physiotherapy in the treatment of osteoarthritis of the hip or knee: protocol of a prospective randomised controlled clinical trial. BMC Musculoskelet Disord. 2009 Aug 19;10:104. doi: 10.1186/1471-2474-10-104. PMID 19689824